CLINICAL TRIAL: NCT01836848
Title: Continuous, Non-invasive Monitoring of Cerebral Oxygenation and Perfusion Using Near-infrared Spectroscopy With Indocyanine Green Perfusion Measurement in Patients With Traumatic Brain Injury, Intracerebral or Subarachnoid Hemorrhage
Brief Title: Non-invasive Measuring of Cerebral Perfusion After Severe Brain Injury With Near-infrared-spectroscopy and ICG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Gerrit Brinker, senior physician, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCH-NIRS-001
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Intracerebral Hemorrhage (ICH); Traumatic Brain Injury
Keywords: subarachnoid hemorrhage; near-infrared-spectroscopy; indocyanine green; secondary ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebral Hemorrhage; Brain Injuries, Traumatic | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- indocyanine green (Experimental): in this arm we do the Intervention 'measuring cerebral perfusion by NIRS with ICG', the pat. gets before a CT-Scan with perfusion measurement a indocyanine green bolus i.v. and a measurement of cerebral perfusion with near-infrared-spectroscopy
  Interventions: Procedure: measuring cerebral perfusion by NIRS with ICG

INTERVENTIONS:
Procedure: measuring cerebral perfusion by NIRS with ICG — application of a bolus of 5mg indocyanine green (ICG) in 3ml saline 0,9% i.v. in 1 second and measuring the ICG turnover with the near-infrared-spectroscopy (NIRS)
  Other Names: indocyanine green; NIRO-200NX C10488, Hamamatsu Photonics K.K.

SUMMARY:
The purpose of this study is to show if it is possible to detect secondary ischemic events in patients with severe brain injury or cerebral haemorrhage with the help of non-invasive near-infrared spectroscopy (NIRS) by using the indocyanine green measuring of cerebral perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* onset of clinical symptoms of subarachnoid or intracranial haemorrhage or trauma suffered less than 72h
* indication for implanting a tissue oxygen and intracranial pressure probe
* A signed informed consent by the patient or legal guardian

Exclusion Criteria:

* Persistent epidural, subdural or subcutaneous hematoma in planned area of the NIRS optode
* Open injuries in the area of the planned optodes
* Malignant primary disease under chemotherapy
* pregnancy
* bleeding disorder
* In the short term unfavorable prognosis (eg, bilateral wide and light-fixed pupils)
* Patients with pacemakers or where no MRI compatibility is due to non- removable metal parts
* contraindications for contrast media in CT (eg, iodine allergy)
* Untreated hyperthyroidism
* End Stage Renal Disease
* severe psychomotor agitation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
with near-infrared-spectroscopy detected cerebral perfusion deficit | 15 days after ictus

SECONDARY OUTCOMES:
Determining a threshold value for cerebral autoregulation measured with near-infrared-spectroscopy as a predictive value for the clinical outcome | 15 days after ictus and follow up 6 month later

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Brinker, physician, Principal Investigator — Universitiy of Cologne, Departement of General Neurosurgery
Locations (1):
- Departement of General Neurosurgery of th University of Cologne, Cologne, Germany